CLINICAL TRIAL: NCT05985733
Title: The Evaluation of Oxidative Stress and Inflammation Markers in Serum and Saliva of the Patients With Temporomandibular Disorders
Brief Title: Evaluation of Oxidative Stress and Inflammation Markers in Temporomandibular Disorders
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Dilara KAZAN, Assistant Professor, Bahçeşehir University
Other Study IDs: PYO.DIS.1904.17.018
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Temporomandibular Disorder; Oxidative Stress; Inflammation
MeSH Terms: conditions — Temporomandibular Joint Disorders; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: patients who applied to our clinic with complaint of pain in TMJ region subjects who had RDC/TMD type II disorder
  Interventions: Other: Biochemical analysis
- Control group: age and sex matched healthy volunteers
  Interventions: Other: Biochemical analysis

INTERVENTIONS:
Other: Biochemical analysis — Oxidative stress and inflammation markers were analyzed in serum and saliva of TMD and healthy subjects.

SUMMARY:
Background: The occurrence of many diseases has been associated with oxidative stress and disruption of antioxidant mechanisms. Temporomandibular Joint(TMJ) Disorders are also thought to develop with the onset of the destructive process in the tissues as a result of this balance being disrupted.

Purpose: This study was designed to compare salivary and serum oxidative stress and inflammation markers of individuals with Temporomandibular Disorders (TMD) and healthy subjects.

Study design, setting, and sample: A prospective cross-sectional study was conducted. 27 TMD patients diagnosed with disc displacement (DD) according to RDC/TMD and 17 healthy subjects were enrolled in the study. Prior to any treatment, serum and saliva samples were taken from the patients and centrifuged, and stored at -80°C until analyzed. All samples were examined for IL-6, MDA and 8-OHdG concentrations.

Predictor variable: Diagnosis of disc displacement (RDC/TMD) Main outcome variables: Levels of 8-OHdG, IL-6 and MDA Covariates: Age and gender

DETAILED DESCRIPTION:
The term oxidative stress is defined as any condition that causes free radical accumulation in tissue. Oxidative stress, which is an indicator of the deterioration of the balance between oxidant/antioxidant in an organism, is thought to play a role in the pathogenesis of various diseases such as atherosclerosis, aging, cancer, neurological disorders, diabetes, ischemia/reperfusion, Alzheimer's, Parkinson's, rheumatoid arthritis and chronic inflammation. Recently, many studies have shown a relationship between the pathogenesis of TMD and various free radicals, antioxidant enzymes and inflammation mediators. Through biomolecule methods studies determine the increase of some of cytokines such as Interleukin 1β (IL-1β), IL-6 in TMJ with internal derangement. These studies emphasize the positive relationship between the severity of the disease and the levels of synovial fluid mediators in joints with TMD. Although it has been supported by previous studies that synovial fluid is a reliable diagnostic material-that reflects the pathological condition in the joint, the disadvantages of the difficulty of obtaining has led to the need for the use of another realiable diagnostic tool. Saliva and blood are materials that are easily available and provide information about the formation and etiology of many systemic diseases.

The aim of this study is to compare the salivary and serum oxidative stress and inflammatory marker levels of TMD patients with RDC/TMD type II disorder with healthy subjects. For this purpose, IL-6, MDA and 8-OHdG will be evaluated as biomarkers of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* TMD subjects who had RDC/TMD type II disorder (TMJ disc displacement (DD) with reduction
* TMJ-DD without reduction with limited opening
* TMJ-DD without reduction without limited opening)

Exclusion Criteria:

* other local or systemic diseases,
* pain of dental origin,
* pregnancy or lactation,
* story of the use of anti-inflammatory drugs, analgesics, muscle relaxants, vitamin C or vitamin E,
* smoking,
* individuals who had already been under treatment for TMD

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: TMD subjects who had RDC/TMD type II disorder (TMJ disc displacement (DD) with reduction, TMJ-DD without reduction with limited opening, TMJ-DD without reduction without limited opening) and, age and sex matched volunteers were included as the control group
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
relationship between serum and salivary 8-OHdG, IL-6 and MDA levels | through study completion, an average of 1 year
  relationship between serum and salivary 8-OHdG, IL-6 and MDA levels and Temporomandibular Disorders were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Dilara Kazan, Principal Investigator — Bahçeşehir University
Locations (1):
- Bahcesehir University, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No